CLINICAL TRIAL: NCT06406868
Title: Effect of Outpatient Versus Tele Rehabilitation on Shoulder Functional Independence Among Post-surgical Breast Cancer Survivors
Brief Title: Outpatient Versus Tele Rehabilitation Among Post-surgical Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01729 Qurat ul ain Khan
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Shoulder Functional Independece
MeSH Terms: conditions — Breast Neoplasms | interventions — American Cancer Society

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehablitation (Experimental): The treatment plan of both groups will be the same according to the exercise plan given by American Cancer Society guidelines for breast cancer patients.
  Frequency :10 repetitions Intensity: Moderate Time: Once a day
  Interventions: Other: American Cancer Society
- Outpatient Rehablitation (Active Comparator): The treatment plan of both groups will be the same according to the exercise plan given by American Cancer Society guidelines for breast cancer patients.
  Frequency :10 repetitions Intensity: Moderate Time: Once a day
  Interventions: Other: American Cancer Society

INTERVENTIONS:
Other: American Cancer Society — After taking base line readings the patients will be divided into two groups' experimental group and control group by randomization. The experimental group will receive tele rehabilitation and the control group will receive outpatient rehabilitation. Readings will be taken at the end of every week. The treatment plan of both groups will be the same according to the exercise plan given by American Cancer Society guidelines for breast cancer patients. The exercise plan will start on third day of surgery. A pictorial reference will be given to every patient to perform exercise.
  The exercise session will be thrice a week, for 60 min, and for four consecutive weeks, for 12 sessions. Exercise plan consists of three phases:
  warm up, balance exercise ,cool down

SUMMARY:
This study is comparing two interventions to identify effective treatment for breast cancer patients.

DETAILED DESCRIPTION:
Tele rehabilitation has gained popularity during Covid 19 pandemic. All the studies carried out at that time was found effective in many countries. Still a literature gap is present in tele rehabilitation in breast cancer patients in Pakistan. Prevalence of breast cancer is high in Pakistan. Now it is the best time to implement tele rehabilitation for breast cancer patients as it will reduce treatment costs and travel expenses. Therefore, the goal of this RCT is to consider tele rehabilitation as part of our treatment plan because if it is found effective for patients than it will be helpful in the field of health and technology.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60 years.
* Breast Cancer Females who underwent mastectomy (Simple total mastectomy).
* Breast Cancer Females without chemotherapy or radiotherapy treatment.
* Accessibility to smart phone.
* Internet access.

Exclusion Criteria:

* Previous history of breast or any other cancer.
* Females with metastatic breast cancer.
* Any Chronic pathology that will result in an increase in symptoms due to physical exercise.
* Any contraindications limiting physical activity.
* Shoulder radiculopathy, or fracture.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast cancer mostly affects females.
Enrollment: 44 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 3rd day
  Changes from baseline are taken shoulder pain disability index is developed to measure shoulder functional independence.It contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. Score ranges from 0 to 100, with higher scores indicating greater shoulder pain and disability.

SECONDARY OUTCOMES:
Breast Cancer Therapy Functional Rating Scale (FACT-B) | 3rd day
  Changes from baseline are taken FACT-B assesses the various domains such as, Physical Well-being, Social/Family Well-being, Emotional Well-being, Functional Well-being, and Additional concerns specific to breast cancer patients.Score ranges from 0 to 148, with 148 a good score
Goniometer | 3rd day
  Changes from baseline ROM of shoulder was taken with the help of goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul ain Khan, MS, Principal Investigator — Riphah International University
Locations (1):
- Nishtar Hospital, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akram M, Iqbal M, Daniyal M, Khan AU. Awareness and current knowledge of breast cancer. Biol Res. 2017 Oct 2;50(1):33. doi: 10.1186/s40659-017-0140-9. PMID 28969709
- [Background] Lee CH, Chung SY, Kim WY, Yang SN. Effect of breast cancer surgery on chest tightness and upper limb dysfunction. Medicine (Baltimore). 2019 May;98(19):e15524. doi: 10.1097/MD.0000000000015524. PMID 31083196
- [Background] Akca M, Ata A, Nayir E, Erdogdu S, Arican A. Impact of Surgery Type on Quality of Life in Breast Cancer Patients. J Breast Health. 2014 Oct 1;10(4):222-228. doi: 10.5152/tjbh.2014.1919. eCollection 2014 Oct. PMID 28331675
- [Background] van Egmond MA, van der Schaaf M, Vredeveld T, Vollenbroek-Hutten MMR, van Berge Henegouwen MI, Klinkenbijl JHG, Engelbert RHH. Effectiveness of physiotherapy with telerehabilitation in surgical patients: a systematic review and meta-analysis. Physiotherapy. 2018 Sep;104(3):277-298. doi: 10.1016/j.physio.2018.04.004. Epub 2018 Jun 19. PMID 30030037
- [Background] Torres-Lacomba M, Sanchez-Sanchez B, Prieto-Gomez V, Pacheco-da-Costa S, Yuste-Sanchez MJ, Navarro-Brazalez B, Gutierrez-Ortega C. Spanish cultural adaptation and validation of the shoulder pain and disability index, and the oxford shoulder score after breast cancer surgery. Health Qual Life Outcomes. 2015 May 23;13:63. doi: 10.1186/s12955-015-0256-y. PMID 26001890
- [Background] Ng R, Lee CF, Wong NS, Luo N, Yap YS, Lo SK, Chia WK, Yee A, Krishna L, Goh C, Cheung YB. Measurement properties of the English and Chinese versions of the Functional Assessment of Cancer Therapy-Breast (FACT-B) in Asian breast cancer patients. Breast Cancer Res Treat. 2012 Jan;131(2):619-25. doi: 10.1007/s10549-011-1764-z. Epub 2011 Sep 16. PMID 21922244
- [Background] Rasmussen GHF, Kristiansen M, Arroyo-Morales M, Voigt M, Madeleine P. Absolute and relative reliability of pain sensitivity and functional outcomes of the affected shoulder among women with pain after breast cancer treatment. PLoS One. 2020 Jun 3;15(6):e0234118. doi: 10.1371/journal.pone.0234118. eCollection 2020. PMID 32492064